CLINICAL TRIAL: NCT00257205
Title: A Phase 3, Open Label, Randomized, Comparative Study Of CP-675,206 And Either Dacarbazine Or Temozolomide In Patients With Advanced Melanoma
Brief Title: CP-675,206 Versus Either Dacarbazine Or Temozolomide In Patients Without Prior Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3671009
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine; tremelimumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Active Comparator): Choice of one or the other Dacarbazine or Temozolomide(CP-675,206) (choice)
  Interventions: Drug: dacarbazine; Drug: temozolomide
- A (Experimental)
  Interventions: Drug: CP-675,206

INTERVENTIONS:
Drug: dacarbazine — decarbazine 1000 mg/m2 IV Q 21 days x 12
  Arms: B
Drug: CP-675,206 — CP-675,206 15 mg/kg IV Q 90 days x 4
  Other Names: anti-CTLA4 human monoclonal antibody
  Arms: A
Drug: temozolomide — temozolomide 200 mg/m2 orally on Days 1-5 every 28 days x 12
  Arms: B

SUMMARY:
This is a Phase 3, multi-national, open-label, 2-arm randomized study in patients with surgically incurable metastatic melanoma who have received no prior chemotherapy, or biochemotherapy for the treatment of metastatic disease. The primary objective of this trial is to compare overall survival for patients with advanced melanoma who are randomized to receive CP-675,206 with that of patients who are randomized to receive either dacarbazine or temozolomide (investigator choice)

ELIGIBILITY:
Inclusion Criteria:

* Surgically incurable melanoma, either Stage IV or IIIC with N3 status for regional lymph nodes and in-transit or satellite lesions.
* Serum lactic acid dehydrogenase (LDH) <= 2 x ULN
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Received any systemic therapy for metastatic melanoma except post-surgical adjuvant treatment with cytokines (eg, alpha-interferon or GM-CSF) or with vaccines after complete resection of melanoma.
* History of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2006-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
overall survival | August 2010

SECONDARY OUTCOMES:
adverse events | 1 year
PFS at 6 months | 6 months
objective tumor response | 1 year
Durable response | 6 months
pharmacokinetics endpoints | 15 months
pharmacogenomic endpoints | 1 year
HQol | 1 year
healthcare resource utilization and loss of productivity | 1 year
human antihuman antibody response for patients in Arm A | 15 months

CONTACTS AND LOCATIONS:
Locations (132):
- United States (48):
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Corona, California
  - Research Site, Fullerton, California
  - Research Site, Glendora, California
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Oxnard, California
  - Research Site, Pasadena, California
  - Research Site, Pomona, California
  - Research Site, Rancho Cucamonga, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Maria, California
  - Research Site, West Covina, California
  - Research Site, Aurora, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Zion, Illinois
  - Research Site, Beech Grove, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Creve Coeur, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Morristown, New Jersey
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dover, Ohio
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Federal Way, Washington
  - Research Site, Lakewood, Washington
  - Research Site, Tacoma, Washington
- Research Site, Ciudad de Buenos Aires, Buenos Aires, Argentina
- Australia (6):
  - Research Site, Waratah, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Woolloongabba, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Launceston, Tasmania
  - Research Site, East Melbourne, Victoria
- Research Site, Vienna, Austria
- Belgium (7):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Namur
  - Research Site, Roeselare
  - Research Site, Turnhout
  - Research Site, Wilrijk
  - Research Site, Yvoir
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (9):
  - Research Site, Montpellier, Cedex 05
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Boulogne
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
- Germany (5):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Tübingen
- Research Site, Athens, Greece
- Israel (3):
  - Research Site, Jerusalem
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (6):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Siena
- Research Site, Mexico City, Mexico City, Mexico
- Netherlands (4):
  - Research Site, Amsterdam, North Holland
  - Research Site, Groningen, Provincie Groningen
  - Research Site, Leiden, South Holland
  - Research Site, Nijmegen
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lubin
  - Research Site, Poznan
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Obninsk, Kaluga Oblast
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Bratislava, Slovakia
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Pretoria
- Spain (8):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Barcelona, Barcelona
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Santander, Cantabria
  - Research Site, Madrid, Madrid
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Zaragoza, Zaragoza
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Lund
- Research Site, Zurich, Switzerland
- United Kingdom (7):
  - Research Site, Truro, Cornwall
  - Research Site, Northwood, Middlesex
  - Research Site, Sutton, Surrey
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Friedlander P, Wood K, Wassmann K, Christenfeld AM, Bhardwaj N, Oh WK. A whole-blood RNA transcript-based gene signature is associated with the development of CTLA-4 blockade-related diarrhea in patients with advanced melanoma treated with the checkpoint inhibitor tremelimumab. J Immunother Cancer. 2018 Sep 18;6(1):90. doi: 10.1186/s40425-018-0408-9. PMID 30227886
- [Derived] Ribas A, Kefford R, Marshall MA, Punt CJ, Haanen JB, Marmol M, Garbe C, Gogas H, Schachter J, Linette G, Lorigan P, Kendra KL, Maio M, Trefzer U, Smylie M, McArthur GA, Dreno B, Nathan PD, Mackiewicz J, Kirkwood JM, Gomez-Navarro J, Huang B, Pavlov D, Hauschild A. Phase III randomized clinical trial comparing tremelimumab with standard-of-care chemotherapy in patients with advanced melanoma. J Clin Oncol. 2013 Feb 10;31(5):616-22. doi: 10.1200/JCO.2012.44.6112. Epub 2013 Jan 7. PMID 23295794